CLINICAL TRIAL: NCT06059326
Title: A Multicenter, Randomized, Double-blind, Placebo Control, Dose-escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of HSK7653 in Type 2 Diabetes Mellitus Patients
Brief Title: Multiple-dose Study to Evaluate the Safety,Tolerability, Pharmacokinetics and Pharmacodynamics of HSK7653 in T2DM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: HSK7653-201
Record Dates: First submitted 2023-09-23; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HSK7653 10 mg (Experimental)
  Interventions: Drug: HSK7653 10 mg
- HSK7653 25 mg (Experimental)
  Interventions: Drug: HSK7653 25 mg
- HSK7653 50 mg (Experimental)
  Interventions: Drug: HSK7653 50 mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HSK7653 10 mg — Tablet, HSK7653 10 mg Q2W, 12 weeks
  Arms: HSK7653 10 mg
Drug: HSK7653 25 mg — Tablet, HSK7653 25 mg Q2W, 12 weeks
  Arms: HSK7653 25 mg
Drug: HSK7653 50 mg — Tablet, HSK7653 50 mg Q2W, 12 weeks
  Arms: HSK7653 50 mg
Drug: Placebo — Tablet, 0 mg Q2W, 12 weeks
  Arms: Placebo

SUMMARY:
To evaluate the safety, tolerability and pharmacokinetic (PK)/pharmacodynamic (PD) characteristics of HSK7653 tablets in Type 2 Diabetes Mellitus Patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 and Age ≤70 years
* T2DM patients,
* Control the blood glucose level only with diet and exercise in last 3 months;
* BMI ≥19 and BMI ≤ 35 kg/m2 (Body Mass Index)
* HbA1c ≥7.0% and HbA1c <10.0%
* FPG <13.9 mmol/L

Exclusion Criteria:

* Non-type 2 diabetes mellitus: Type 1 diabetes mellitus, gestational diabetes history;
* History of acute complications of diabetes (diabetic ketoacidosis, diabetic hyperglycemia hyperosmolar syndrome or lactic acidosis);
* History of chronic complications of severe diabetes (retinal proliferative disease, severe diabetic neuropathy or intermittent claudication confirmed by fundus examination during screening);
* Patients who used systemic glucocorticoids within 3 months prior to screening had severe infections or major surgeries and transplants within 3 months;
* Three or more episodes of hypoglycemia occurred in the six months prior to screening;
* History of hyperthyroidism within 6 months before screening;
* Severe cardiovascular disease. ;
* Medical conditions that may significantly affect drug absorption, distribution, metabolism, and excretion within 2 weeks prior to screening;
* Liver function tests abnormal;
* Moderate or severe renal impairment;
* Medical history or clinical evidence of pancreatic injury or pancreatitis, or abnormalities in lipase and amylase judged by investigators to be clinically significant;
* Patients with a history of hypertension who regularly take antihypertensive therapy for over 4 weeks still have poor control, SBP > 160 mmHg and (or) DBP > 100 mmHg;
* Patients with uncontrolled hyperlipidemia.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-01-22 (Actual); Primary Completion 2019-11-05 (Actual); Study Completion 2019-11-05 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Emergent Adverse Events (TEAEs) | From baseline to up to 2 weeks after last dose for a total of approximately 14 weeks
  Assessment by adverse event monitoring, 12 lead ECGs, vital signs and laboratory measurements.

SECONDARY OUTCOMES:
Peak plasma concentration (Cmax) of HSK7653 | Day 1 to Day 43
  Cmax of HSK7653 after first dose and multi-dose administration
Area under the plasma concentration versus time curve (AUC) of HSK7653 | Day 1 to Day 43
  AUC of HSK7653 after first dose and multi-dose administration
Half-life (t1/2) of HSK7653 | Day 1 to Day 43
  T1/2 of HSK7653 after single-dose and multi-dose administration
Change from baseline in dipeptidyl peptidase-IV (DPP-4) inhibition rate | Day 1 to Day 84
  Change from baseline in dipeptidyl peptidase-IV (DPP-4) inhibition rate after single-dose and multi-dose administration of HSK7653
Change from baseline in GLP-1 | Day 1 to Day 84
  Change from baseline in GLP-1 after single-dose and multi-dose administration of HSK7653
Change from baseline of fasting plasma glucose | Day 1 to Day 84
  Change from baseline in fasting plasma glucose after multi-dose administration of HSK7653
Change from baseline of HbA1c | Day 1 to Day 84
  Change from baseline in HbA1c after multi-dose administration of HSK7653

CONTACTS AND LOCATIONS:
Locations (1):
- Peking university people's hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No